CLINICAL TRIAL: NCT03530774
Title: Egg Protein Supplementation for Maintaining Muscle Mass and Function in Older Adults
Brief Title: Supplemental Egg Protein Intervention in Older Adults
Acronym: SPRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at San Antonio (Other)
Collaborators: Texas State University (Other); American Egg Board (Other)
Responsible Party: Principal Investigator, Sarah Ullevig, Assistant Professor, The University of Texas at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 17-110
Record Dates: First submitted 2017-10-13; First posted 2018-05-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2020-11

CONDITIONS: Sarcopenia; Aging
Keywords: physical performance battery; 24-hour dietary recalls; dual-energy X-ray absorptimetry; dietary supplement; protein
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to control (carbohydrate) or egg white protein supplement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Egg while protein supplement (Experimental): 25 g of powdered egg white protein supplement daily for 6 months. Total of 20.6 g of protein in 25 g of supplement.
  Interventions: Dietary Supplement: powdered egg white protein supplement
- Maltodextrin supplement (Placebo Comparator): 25 g of powdered maltodextrin supplement daily for 6 months. Total 23.5 g of carbohydrate in 25 g of supplement.
  Interventions: Dietary Supplement: maltodextrin supplement

INTERVENTIONS:
Dietary Supplement: powdered egg white protein supplement — consumption of egg white protein supplement daily for 6 months
  Arms: Egg while protein supplement
Dietary Supplement: maltodextrin supplement — consumption of maltodextrin supplement daily for 6 months
  Arms: Maltodextrin supplement

SUMMARY:
Older adults are at risk for developing sarcopenia, or age-related muscle loss, which increased the risk of disabilities, falls, and loss of independence. Many older adults do not consume enough protein each day to maintain their muscle mass and this study aims to investigate if consumption daily egg white protein supplement can help maintain muscle mass and functionality in community-dwelling older adults. Food insecure older adults that attend congregate nutrition sites will be targeted.

DETAILED DESCRIPTION:
The study aims to evaluate the impact of egg white protein supplementation on muscle mass, strength, and physical function in older adults with low muscle mass or function. Older adults will be recruited from San Antonio, Texas, the least food secure metropolitan area for older adults. The project will be conducted entirely at community locations such as congregate meal sites, senior activity centers, and housing communities. Researchers will conduct recruitment, distribution of supplements and pre and post assessments entirely at these sites, which will alleviate the travel of participants to research sites and provide a unique opportunity to assess this underserved population. One hundred older adults (≥60yrs old) will be randomly assigned to consume a daily supplement of egg white protein or isoenergetic carbohydrate for 6 months. Changes in skeletal muscle mass, muscle strength, and physical function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older, gait speed >0.8m/s OR hand grip below 20kg for women or below 30kg for men

Exclusion Criteria:

* Over 300 pounds, kidney disease, has taken a protein supplement within the past 30 days, dementia/Alzheimer's, uncontrolled diabetes, wheelchair bound, vegan, allergic to eggs, blind/legally blind, history of stroke/transient ischemic attack with a Barthel score of 15 or lower, cannot read or write English or Spanish and don't have someone to help them with forms/paperwork, not willing to take a supplement for 6 months or will not remain in the local area for the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Muscle mass | Change from Baseline Muscle Mass at 6 months
  Dual-energy X-ray absorptimetry
Short physical performance battery (SPPB) | Change from Baseline Physical Function at 6 months
  Includes objective, performance-based measures of balance (standing side by side, semi-tandem and tandem), mobility (4-m habitual gait speed), and strength (5 chair stands). Each task is scored from 0-4 Points (p) and then summed into a total score of 0 (worst)-12 (best) p, where 12 p represents the highest performance.
Muscle Strength | Change from Baseline Muscle Strength at 6 months
  Hand Dynamometer

SECONDARY OUTCOMES:
Protein intake | Change from Baseline Protein Intake at 6 months
  24-hour recalls (2 non-consecutive)
Health-Related Quality of Life | Change from Baseline Health-Related Quality of Life at 6 months
  Short Form 12 Health Survey
Upper Respiratory Illnesses Frequency | Change From Baseline Upper Respiratory Illness Frequency at 6 months
  Daily illness log
Cognitive Function | Change from Baseline Cognitive Function at 6 months
  Trail Making Test A and B
Falls Risk | Change From Baseline Falls Efficacy and Frequency at 6 months
  A short questionnaire will be used to gather information on number of falls recalled over the past 6 months, whether the individual sought medical attention for any of the falls, and whether an injury resulted from any of the falls. The Falls Efficacy Scale is a 10 item scale assessing the confidence level individuals have in performing daily activities without falling. Each item is rated on a scale of 0-10, with 0 signifying no confidence and 10 indicating very confident. Scores are totaled and range from 0-100 with higher scores indicating greater confidence
Functional Limitations and Disability | Change From Baseline Functional Limitations and Disability at 6 months
  The Late-Life Function and Disability Instrument is a validated questionnaire that measures both functional limitations and disability. The function component evaluates self-reported difficulty in performing 32 physical activities. Scores range from 0-100 with higher scores indicating higher levels of function. Disability component evaluates self-reported limitations and frequency of limitations in 16 activities. Scores range from 0-100 with higher scores indicating higher levels of function.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Ullevig, PhD, RD, Principal Investigator — University of Texas at San Antonio
Locations (1):
- University of Texas at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Drewnowski A, Specter SE. Poverty and obesity: the role of energy density and energy costs. Am J Clin Nutr. 2004 Jan;79(1):6-16. doi: 10.1093/ajcn/79.1.6. PMID 14684391
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Janssen I, Shepard DS, Katzmarzyk PT, Roubenoff R. The healthcare costs of sarcopenia in the United States. J Am Geriatr Soc. 2004 Jan;52(1):80-5. doi: 10.1111/j.1532-5415.2004.52014.x. PMID 14687319
- [Background] Ali S, Garcia JM. Sarcopenia, cachexia and aging: diagnosis, mechanisms and therapeutic options - a mini-review. Gerontology. 2014;60(4):294-305. doi: 10.1159/000356760. Epub 2014 Apr 8. PMID 24731978
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753
- [Background] Best RL, Appleton KM. The consumption of protein-rich foods in older adults: an exploratory focus group study. J Nutr Educ Behav. 2013 Nov-Dec;45(6):751-5. doi: 10.1016/j.jneb.2013.03.008. Epub 2013 Jul 2. PMID 23827439
- [Background] Paddon-Jones D, Rasmussen BB. Dietary protein recommendations and the prevention of sarcopenia. Curr Opin Clin Nutr Metab Care. 2009 Jan;12(1):86-90. doi: 10.1097/MCO.0b013e32831cef8b. PMID 19057193
- [Background] Lloyd JL, Wellman NS. Older Americans Act Nutrition Programs: A Community-Based Nutrition Program Helping Older Adults Remain at Home. J Nutr Gerontol Geriatr. 2015;34(2):90-109. doi: 10.1080/21551197.2015.1031592. PMID 26106983
- [Background] Milne AC, Avenell A, Potter J. Meta-analysis: protein and energy supplementation in older people. Ann Intern Med. 2006 Jan 3;144(1):37-48. doi: 10.7326/0003-4819-144-1-200601030-00008. PMID 16389253
- [Derived] Ullevig SL, Zuniga K, Austin Lobitz C, Santoyo A, Yin Z. Egg protein supplementation improved upper body muscle strength and protein intake in community-dwelling older adult females who attended congregate meal sites or adult learning centers: A pilot randomized controlled trial. Nutr Health. 2022 Dec;28(4):611-620. doi: 10.1177/02601060211051592. Epub 2021 Nov 3. PMID 34730461
- See also: Ziliak JP, Gundersen C. The Health Consequences of Senior Hunger in the United States : Evidence from the 1999-2010 NHANES. 2014. — https://www.feedingamerica.org/sites/default/files/research/senior-hunger-research/senior-health-consequences-2014.pdf
- See also: Borger C, Dys TD, Engelhard E, et al. Hunger in America 2014: Executive summary. 2014 — http://help.feedingamerica.org/HungerInAmerica/hunger-in-america-2014-summary.pdf
- See also: Strickhouser S, Wright JD, Donley AM. Food insecurity among older adults. AARP Foundation. 2015. — http://www.aarp.org/content/dam/aarp/aarp_foundation/2015-PDFs/AF-Food-Insecurity-2015Update-Final-Report.pdf